CLINICAL TRIAL: NCT01667055
Title: The Optimized Diagnostic Methods for the Confirmation of Beta-lactam Hypersensitivity in Thailand
Brief Title: The Diagnosis of Beta-lactam Hypersensitivity in Thailand
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Jettanong Klaewsongkram, MD., Associate Professor, Chulalongkorn University
Other Study IDs: Chula-ARC 002/12
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Penicillin Allergy; Aminopenicillin Allergy; Beta Lactam Adverse Reaction
Keywords: drug allergy; drug hypersensitivity; beta-lactam allergy; penicillin allergy; adverse drug reaction
MeSH Terms: conditions — Drug Hypersensitivity; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells in patients with a history of non-immediate reaction
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with suspected drug allergy: Patients with a history of hypersensitivity reaction to beta-lactam antibiotics

SUMMARY:
The true prevalence of drug allergy in patients with a history of beta-lactam hypersensitivity will be determined by using commercially available standard skin test reagents and the diagnostic agents available in Thailand. We hypothesize that only minority of patients with such a history are truly allergic.

DETAILED DESCRIPTION:
Patients with a history of beta-lactam hypersensitivity will be evaluated by the standard skin test reagents (major and minor determinants of penicillin, amoxicillin, and clavulanic if applicable), and intravenous forms of beta-lactam antibiotics .

Diagnostic values of the measurement of specific Immunoglobulin E to penicillin/aminopenicillin and skin test reagents currently available in Thailand will be comparatively analyzed with the standard skin test reagents.

The measurement of drug-induced interferon-gamma releasing cells will be measured in patients with a history of non-immediate reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of beta-lactam hypersensitivity

Exclusion Criteria:

* Being pregnant
* Having serious medical illnesses

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a history of beta-lactam hypersensitivity
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The true prevalence of drug allergy in patients with a history of beta-lactam hypersensitivity | 1 year
  The skin test positive rate in patients with a history of beta-lactam hypersensitivity

SECONDARY OUTCOMES:
Clinical values of various diagnostic modalities in patients with a history of beta-lactam hypersensitivity | 1 year
  The diagnostic values of skin testing, drug-specific Immunoglobulin E measurement, and interferon-gamma ELISpot assay for the diagnosis of beta-lactam hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chongpison Y, Palapinyo S, Mongkolpathumrat P, Buranapraditkun S, Thantiworasit P, Klaewsongkram J. Beta-lactam hypersensitivity diagnosis in ambulatory and hospitalized settings require different approaches. Ann Allergy Asthma Immunol. 2023 Jan;130(1):84-92.e1. doi: 10.1016/j.anai.2022.09.011. Epub 2022 Sep 16. PMID 36122888